CLINICAL TRIAL: NCT01338545
Title: A Multi-centre Observational Study to Describe Usage and Dosification Patterns of RoActemra (Tocilizumab) Treatment in Rheumatoid Arthritis (RA) Patients in the Routine Clinical Practice. ACT-LIFE Study
Brief Title: An Observational Study of Dosage Patterns in Routine Clinical Practice in Patients With Rheumatoid Arthritis (ACT-LIFE)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25264
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the dosage patterns, safety and efficacy of RoActemra/Actemra (tocilizumab) in clinical practice in patients with moderate to severe rheumatoid arthritis who have not responded or are intolerant to at least one disease-modifying antirheumatic drug (DMARD) or TNF inhibitor. Data will be collected from each patients for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis (RA) of at least 6 months duration
* Non-responder or intolerant to at least one DMARD or TNF inhibitor treatment
* Initiated on treatment with RoActemra according to Summary of Product Characteristics (SPC) indications

Exclusion Criteria:

* History of autoimmune disease or of any joint inflammatory disease other than RA
* Pregnant or lactating women
* Patients who have started RoActemra treatment in a clinical trial or for compassionate use
* Treatment with any investigational drug in the previous 4 weeks (or at least 5 times the half-life of the drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis initiated on treatment with RoActemra/Actemra after at least one previous DMARD or TNF-inhibitor treatment
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Changes in treatment schedules (dosage reduction/interruption/discontinuation) for safety reasons | 12 months

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | 12 months
Change in disease activity (disease activity score DAS28/ simple disease activity index SDAI) | 12 months
Response rate according to EULAR (European League Against Rheumatism) criteria | 12 months
Quality of life (Visual Analogue Scales, Health Assessment Questionnaire) | 12 months
Response/tolerance with regard to pretreatment with either DMARDs or TNF inhibitors | 12 months
Effect on DMARD tolerance/dosage in combination therapy | 12 months
Dosages used in clinical practice | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- Coral Springs, Florida, United States
- Spain (38):
  - Elche, Alicante
  - Elda, Alicante
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Sant Joan Despí, Barcelona
  - Jerez de la Frontera, Cadiz
  - Santander, Cantabria
  - Torrelavega, Cantabria
  - Castellon, Castellon
  - Vinaròs, Castellon
  - Córdoba, Cordoba
  - Girona, Girona
  - Granada, Granada
  - Donostia / San Sebastian, Guipuzcoa
  - Huelva, Huelva
  - A Coruña, La Coruña
  - Santiago de Compostela, La Coruña
  - Logroño, La Rioja
  - Alcalá de Henares, Madrid
  - Alcorcón, Madrid
  - El Escorial, Madrid
  - Madrid, Madrid
  - Málaga, Malaga
  - Cartagena, Murcia
  - El Palmar, Murcia
  - Lorca, Murcia
  - Murcia, Murcia
  - Pamplona, Navarre
  - Ourense, Orense
  - Vigo, Pontevedra
  - Seville, Sevilla
  - Toledo, Toledo
  - Alzira, Valencia
  - San Juan, Valencia
  - Valencia, Valencia
  - Valenica, Valencia
  - Barakaldo, Vizcaya
  - Bilbao, Vizcaya